CLINICAL TRIAL: NCT03619213
Title: An International, Double-blind, Randomised, Placebo-Controlled Phase III Study to Evaluate the Effect of Dapagliflozin on Reducing CV Death or Worsening Heart Failure in Patients With Heart Failure With Preserved Ejection Fraction (HFpEF)
Brief Title: Dapagliflozin Evaluation to Improve the LIVEs of Patients With PReserved Ejection Fraction Heart Failure.
Acronym: DELIVER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D169CC00001; 2018-000802-46 (EudraCT Number)
Record Dates: First submitted 2018-08-02; First posted 2018-08-07 (Actual); Results first posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Heart Failure With Preserved Ejection Fraction
MeSH Terms: interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: International, Double-blind, Randomised, Placebo-Controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin (Experimental): Patients will be randomized 1:1 to either dapagliflozin or placebo.
  Interventions: Drug: Dapagliflozin
- Placebo (Placebo Comparator): Placebo matching dapagliflozin.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — 10 mg tablets given once daily, per oral use.
  Other Names: Forxiga TM; Farxiga TM
  Arms: Dapagliflozin
Drug: Placebo — Placebo matching dapagliflozin 10 mg
  Arms: Placebo

SUMMARY:
This is an international, multicentre, parallel-group, event-driven, randomised, double-blind, placebo-controlled study in HFpEF patients, evaluating the effect of dapagliflozin 10 mg versus placebo, given once daily in addition to background regional standard of care therapy, including treatments to control co-morbidities, in reducing the composite of CV death or heart failure events.

DETAILED DESCRIPTION:
This is an international, multicentre, parallel-group, event-driven, randomised, double-blind study in patients with HFpEF, evaluating the effect of dapagliflozin 10 mg versus placebo, given once daily in addition to background regional standard of care therapy, including treatments to control co-morbidities, in reducing the composite of CV death and heart failure events (hospitalisations for HF or urgent HF visits). Adult patients aged ≥40 years with HFpEF (LVEF >40% and evidence of structural heart disease) and New York Heart Association (NYHA) class II-IV who are eligible according to the inclusion/exclusion criteria will be randomised in a 1:1 ratio to receive either dapagliflozin 10 mg or placebo. Both out-patients and in-patients hospitalised for heart failure and off intravenous heart failure-therapy for 24 hours can be randomised. It is estimated that approximately 11000 patients at approximately 400-500 sites in 20-25 countries will need to be enrolled to reach the target of approximately 6100 randomised patients.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed informed consent prior to any study specific procedures.
2. Male or female patients age ≥40 years.
3. Documented diagnosis of symptomatic heart failure (NYHA class II-IV) at enrolment, and a medical history of typical symptoms/signs of heart failure ≥6 weeks before enrolment with at least intermittent need for diuretic treatment.
4. Left Ventricular Ejection Fraction (LVEF) >40% and evidence of structural heart disease (i.e. left ventricular hypertrophy or left atrial enlargement ) documented by the most recent echocardiogram, and/or cardiac MR within the last 12 months prior to enrolment. For patients with prior acute cardiac events or procedures that may reduce LVEF, e.g. as defined in exclusion criterion 6, qualifying cardiac imaging assessment at least 12 weeks following the procedure/event is required.
5. Elevated NT-pro BNP levels.
6. Both ambulatory and hospitalised patients may be enrolled and randomised. Patients currently hospitalised for HF, must be off intravenous HF medications for at least 24 before randomisation.

Further details regarding inclusion criteria 4-6 may apply.

Exclusion Criteria:

1. Receiving therapy with an SGLT2 inhibitor within 4 weeks prior to randomisation or previous intolerance to an SGLT2 inhibitor.
2. Type 1 diabetes mellitus (T1D).
3. eGFR <25 mL/min/1.73 m2 (CKD-EPI formula) at Visit 1.
4. Systolic blood pressure (BP) <95 mmHg on 2 consecutive measurements at 5-minute intervals, at Visit 1 or at Visit 2.
5. Systolic BP≥160 mmHg if not on treatment with ≥3 blood pressure lowering medications or ≥180 mmHg irrespective of treatments, on 2 consecutive measurements at 5-minute intervals, at Visit 1 or at Visit 2.
6. MI, unstable angina, coronary revascularization (percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG)), ablation of atrial flutter/fibrillation, valve repair/replacement within 12 weeks prior to enrolment. Before enrolment, these patients must have their qualifying echocardiography and/or cardiac MRI examination at least 12 weeks after the event.
7. Planned coronary revascularization, ablation of atrial flutter/fibrillation and valve repair/replacement.
8. Stroke or transient ischemic attack (TIA) within 12 weeks prior to enrolment.
9. Probable alternative or concomitant diagnoses which in the opinion of the investigator could account for the patient's HF symptoms and signs (e.g. anaemia, hypothyroidism).
10. Body mass index >50 kg/m2.

Further exclusion criteria may apply

Ages: 40 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6263 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2022-03-27 (Actual); Study Completion 2022-03-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (274):
- United States (60):
  - Research Site, Fairhope, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Sheffield, Alabama
  - Research Site, Tucson, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Beverly Hills, California
  - Research Site, Loma Linda, California
  - Research Site, Los Angeles, California
  - Research Site, Stamford, Connecticut
  - Research Site, Clearwater, Florida
  - Research Site, Miami, Florida
  - Research Site, Naples, Florida
  - Research Site, Ocala, Florida
  - Research Site, Ormond Beach, Florida
  - Research Site, Port Charlotte, Florida
  - Research Site, Saint Augustine, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Gurnee, Illinois
  - Research Site, Anderson, Indiana
  - Research Site, Munster, Indiana
  - Research Site, Louisville, Kentucky
  - Research Site, Hammond, Louisiana
  - Research Site, Houma, Louisiana
  - Research Site, Monroe, Louisiana
  - Research Site, Boston, Massachusetts
  - Research Site, Bay City, Michigan
  - Research Site, Flint, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Rochester, Minnesota
  - Research Site, Saint Paul, Minnesota
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Great Falls, Montana
  - Research Site, Las Vegas, Nevada
  - Research Site, Lebanon, New Hampshire
  - Research Site, Bridgewater, New Jersey
  - Research Site, Buffalo, New York
  - Research Site, New York, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Altoona, Pennsylvania
  - Research Site, Doylestown, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site, Charleston, South Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, Jackson, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Tullahoma, Tennessee
  - Research Site, Beaumont, Texas
  - Research Site, Humble, Texas
  - Research Site, Sherman, Texas
  - Research Site, Burlington, Vermont
  - Research Site, Falls Church, Virginia
  - Research Site, Leesburg, Virginia
  - Research Site, Morgantown, West Virginia
  - Research Site, Madison, Wisconsin
  - Research Site, Milwaukee, Wisconsin
- Argentina (12):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Catamarca
  - Research Site, Ciudad Autonoma de Buenos Aire
  - Research Site, Corrientes
  - Research Site, Córdoba
  - Research Site, Mar del Plata
  - Research Site, Ramos Mejía
  - Research Site, Rosario
  - Research Site, San Miguel de Tucumán
  - Research Site, San Nicolás
  - Research Site, Santa Fe
- Belgium (6):
  - Research Site, Aalst
  - Research Site, Brasschaat
  - Research Site, Brussels
  - Research Site, Huy
  - Research Site, Kortrijk
  - Research Site, Leuven
- Brazil (10):
  - Research Site, Belo Horizonte
  - Research Site, Blumenau
  - Research Site, Campina Grande do Sul
  - Research Site, Campinas
  - Research Site, Curitiba
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, Santo André
  - Research Site, São Paulo
  - Research Site, Votuporanga
- Bulgaria (8):
  - Research Site, Dimitrovgrad
  - Research Site, Haskovo
  - Research Site, Kozloduy
  - Research Site, Pazardzhik
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Sofia
  - Research Site, Stara Zagora
- Canada (18):
  - Research Site, Winnipeg, Manitoba
  - Research Site, Brampton, Ontario
  - Research Site, Burlington, Ontario
  - Research Site, Cambridge, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, North York, Ontario
  - Research Site, Oshawa, Ontario
  - Research Site, Port Perry, Ontario
  - Research Site, Scarborough Village, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Waterloo, Ontario
  - Research Site, York, Ontario
  - Research Site, Laval, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Saint-Jérôme, Quebec
  - Research Site, Terrebonne, Quebec
  - Research Site, Trois-Rivières, Quebec
- China (22):
  - Research Site, Baotou
  - Research Site, Beijing
  - Research Site, Cangzhou
  - Research Site, Changchun
  - Research Site, Chengdu
  - Research Site, Chifeng
  - Research Site, Dalian
  - Research Site, Daqing
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Haerbin
  - Research Site, Jinan
  - Research Site, Lanzhou
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Pingxiang
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Tianjin
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Yinchuan
- Czechia (11):
  - Research Site, Benešov
  - Research Site, Brandýs nad Labem
  - Research Site, Brno
  - Research Site, Jaroměř
  - Research Site, Kladno
  - Research Site, Louny
  - Research Site, Náchod
  - Research Site, Ostrava-Dubina
  - Research Site, Pardubice
  - Research Site, Prague
  - Research Site, Příbram
- Hungary (10):
  - Research Site, Budapest
  - Research Site, Győr
  - Research Site, Kecskemét
  - Research Site, Miskolc
  - Research Site, Nyíregyháza
  - Research Site, Szekszárd
  - Research Site, Szentes
  - Research Site, Székesfehérvár
  - Research Site, Szolnok
  - Research Site, Zalaegerszeg
- Japan (42):
  - Research Site, Adachi-ku
  - Research Site, Asahi-shi
  - Research Site, Azumino-shi
  - Research Site, Beppu-shi
  - Research Site, Chūōku
  - Research Site, Fujisawa-shi
  - Research Site, Funabashi-shi
  - Research Site, Hachioji-shi
  - Research Site, Hamada-shi
  - Research Site, Hamamatsu
  - Research Site, Higashiohmi-shi
  - Research Site, Ichinomiya-shi
  - Research Site, Iizuka-shi
  - Research Site, Iwakuni-shi
  - Research Site, Kanazawa
  - Research Site, Kasugai-shi
  - Research Site, Kawasaki-shi
  - Research Site, Kishiwada-shi
  - Research Site, Kobe
  - Research Site, Koga-shi
  - Research Site, Kuki-shi
  - Research Site, Kure-shi
  - Research Site, Kyoto
  - Research Site, Matsumoto-shi
  - Research Site, Mito
  - Research Site, Miura-gun
  - Research Site, Nakagami-gun
  - Research Site, Nishinomiya-shi
  - Research Site, Ōita
  - Research Site, Saga
  - Research Site, Sagamihara-shi
  - Research Site, Sapporo
  - Research Site, Shinagawa-ku
  - Research Site, Suita-shi
  - Research Site, Takamatsu
  - Research Site, Takasago-shi
  - Research Site, Toride-shi
  - Research Site, Tsu
  - Research Site, Tsuchiura-shi
  - Research Site, Ueda-shi
  - Research Site, Ureshino-shi
  - Research Site, Utsunomiya
- Mexico (10):
  - Research Site, Aguascalientes
  - Research Site, Culiacán
  - Research Site, Guadalajara
  - Research Site, Mazatlán
  - Research Site, México
  - Research Site, Monclova
  - Research Site, Monterrey
  - Research Site, Querétaro
  - Research Site, Tijuana
  - Research Site, Veracruz
- Netherlands (11):
  - Research Site, Amsterdam
  - Research Site, Arnhem
  - Research Site, Dordrecht
  - Research Site, Groningen
  - Research Site, Heerlen
  - Research Site, Leiderdorp
  - Research Site, Meppel
  - Research Site, Rotterdam
  - Research Site, The Hague
  - Research Site, Uden
  - Research Site, Veldhoven
- Peru (7):
  - Research Site, Bellavista
  - Research Site, Callao
  - Research Site, Chancay
  - Research Site, Chorrillos
  - Research Site, Lima
  - Research Site, San Isidro
  - Research Site, Urb. El Chipe
- Poland (16):
  - Research Site, Bialystok
  - Research Site, Bochnia
  - Research Site, Chojnice
  - Research Site, Gdansk
  - Research Site, Gdynia
  - Research Site, Jasło
  - Research Site, Katowice
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Opole
  - Research Site, Oława
  - Research Site, Płock
  - Research Site, Rzeszów
  - Research Site, Torun
  - Research Site, Wierzchosławice
  - Research Site, Wroclaw
- Romania (4):
  - Research Site, Brasov
  - Research Site, Craiova
  - Research Site, Iași
  - Research Site, Tg Mures
- Russia (7):
  - Research Site, Chelyabinsk
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Perm
  - Research Site, Ryazan
  - Research Site, Saint Petersburg
  - Research Site, Tver'
- Saudi Arabia (3):
  - Research Site, Dammam
  - Research Site, Jeddah
  - Research Site, Riyadh
- Spain (9):
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, Hospitalet de Llobregat(Barcel
  - Research Site, Madrid
  - Research Site, Sanlúcar de Barrameda (Cádiz)
  - Research Site, Santiago(A Coruña)
  - Research Site, Seville
  - Research Site, Valencia
  - Research Site, Villamartín (Cádiz)
- Taiwan (6):
  - Research Site, Hsinchu
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan
- Vietnam (2):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Myte R, Mattsson A, Poole M, Little DJ, Nystrom P, Henderson A, Claggett BL, Gasparyan SB, Solomon SD, McMurray JJV. Survival Odds to Minimize Risk Heterogeneity Bias in Heart Failure Trials: Application to Dapagliflozin. Circ Heart Fail. 2025 Dec;18(12):e013496. doi: 10.1161/CIRCHEARTFAILURE.125.013496. Epub 2025 Oct 31. PMID 41170566
- [Derived] Ostrominski JW, Neuen BL, Claggett BL, Anand IS, Desai AS, Jhund PS, Lam CSP, Pfeffer MA, Pitt B, Zannad F, Zile MR, Packer M, Docherty KF, McMurray JJV, Solomon SD, Vaduganathan M. Natriuretic Peptides, Body Mass Index, and Clinical Outcomes in Heart Failure With Mildly Reduced or Preserved Ejection Fraction. J Am Coll Cardiol. 2025 Nov 18;86(20):1823-1839. doi: 10.1016/j.jacc.2025.08.028. Epub 2025 Aug 27. PMID 40892613
- [Derived] Siqueira SRO, Pabon MA, Vaduganathan M, Claggett BL, Lam CSP, Kosiborod MN, de Boer RA, Shah SJ, Fang JC, Desai AS, Jhund PS, Inzucchi SE, Martinez F, Hernandez AF, Petersson M, McMurray JJV, Solomon SD, Vardeny O. Achieved Ejection Fraction and Effects of Dapagliflozin in Heart Failure With Improved Ejection Fraction. JACC Heart Fail. 2025 Oct;13(10):102585. doi: 10.1016/j.jchf.2025.102585. Epub 2025 Aug 19. PMID 40834567
- [Derived] Inciardi RM, Lu H, Claggett BL, Desai AS, Jhund PS, Lam CSP, Kosiborod MN, Inzucchi SE, Martinez FA, de Boer RA, Hernandez AF, Shah SJ, Kober L, Ponikowski P, Sabatine MS, Petersson M, Langkilde AM, McMurray JJV, Vaduganathan M, Solomon SD. Severe Heart Failure and Treatment With Dapagliflozin Across the Ejection Fraction Spectrum: DAPA-HF and DELIVER. JACC Heart Fail. 2025 Apr;13(4):618-627. doi: 10.1016/j.jchf.2024.11.023. Epub 2025 Mar 5. PMID 40047763
- [Derived] Yang M, Kondo T, Talebi A, Jhund PS, Docherty KF, Claggett BL, Vaduganathan M, Bachus E, Hernandez AF, Lam CSP, Martinez FA, de Boer RA, Kosiborod MN, Desai AS, Kober L, Ponikowski P, Sabatine MS, Solomon SD, McMurray JJV. EuroQol 5-Dimension Questionnaire in Heart Failure With Reduced, Mildly Reduced, and Preserved Ejection Fraction: A Patient-Level Analysis of DAPA-HF and DELIVER. JACC Heart Fail. 2025 Feb;13(2):277-292. doi: 10.1016/j.jchf.2024.10.020. PMID 39909641
- [Derived] Lu H, Kondo T, Claggett BL, Vaduganathan M, Neuen BL, Beldhuis IE, Jhund PS, Mc Causland FR, Anand IS, Pfeffer MA, Pitt B, Zannad F, Zile MR, McMurray JJV, Solomon SD, Desai AS. Systolic Blood Pressure and Pulse Pressure in Heart Failure: Pooled Participant-Level Analysis of 4 Trials. J Am Coll Cardiol. 2025 Feb 25;85(7):710-722. doi: 10.1016/j.jacc.2024.11.007. Epub 2024 Nov 15. PMID 39745404
- [Derived] Kondo T, Gasparyan SB, Jhund PS, Bengtsson O, Claggett BL, de Boer RA, Hernandez AF, Inzucchi SE, Kosiborod MN, Kober L, Lam CSP, Langkilde AM, Martinez FA, Petersson M, Ponikowski P, Sabatine MS, Shah SJ, Sjostrand M, Wilderang U, Vaduganathan M, Solomon SD, McMurray JJV. Use of Win Statistics to Analyze Outcomes in the DAPA-HF and DELIVER Trials. NEJM Evid. 2023 Nov;2(11):EVIDoa2300042. doi: 10.1056/EVIDoa2300042. Epub 2023 Oct 24. PMID 38320525
- [Derived] Vardeny O, Desai AS, Jhund PS, Fang JC, Claggett B, de Boer RA, Hernandez AF, Inzucchi SE, Kosiborod MN, Lam CSP, Martinez FA, Shah SJ, Mc Causland FR, Petrie MC, Vaduganathan M, McMurray JJV, Solomon SD. Dapagliflozin and Mode of Death in Heart Failure With Improved Ejection Fraction: A Post Hoc Analysis of the DELIVER Trial. JAMA Cardiol. 2024 Mar 1;9(3):283-289. doi: 10.1001/jamacardio.2023.5318. PMID 38265835
- [Derived] Mc Causland FR, Claggett BL, Vaduganathan M, Desai A, Jhund P, Vardeny O, Fang JC, de Boer RA, Docherty KF, Hernandez AF, Inzucchi SE, Kosiborod MN, Lam CSP, Martinez F, Saraiva JFK, McGrath MM, Shah SJ, Verma S, Langkilde AM, Petersson M, McMurray JJV, Solomon SD. Decline in Estimated Glomerular Filtration Rate After Dapagliflozin in Heart Failure With Mildly Reduced or Preserved Ejection Fraction: A Prespecified Secondary Analysis of the DELIVER Randomized Clinical Trial. JAMA Cardiol. 2024 Feb 1;9(2):144-152. doi: 10.1001/jamacardio.2023.4664. PMID 37952176
- [Derived] Kondo T, Butt JH, Curtain JP, Jhund PS, Docherty KF, Claggett BL, Vaduganathan M, Bachus E, Hernandez AF, Lam CSP, Inzucchi SE, Martinez FA, de Boer RA, Kosiborod MN, Desai AS, Kober L, Ponikowski P, Sabatine MS, Solomon SD, McMurray JJV. Efficacy of Dapagliflozin According to Heart Rate: A Patient-Level Pooled Analysis of DAPA-HF and DELIVER. Circ Heart Fail. 2023 Dec;16(12):e010898. doi: 10.1161/CIRCHEARTFAILURE.123.010898. Epub 2023 Oct 27. PMID 37886880
- [Derived] Ostrominski JW, Vaduganathan M, Selvaraj S, Claggett BL, Miao ZM, Desai AS, Jhund PS, Kosiborod MN, Lam CSP, Inzucchi SE, Martinez FA, de Boer RA, Hernandez AF, Shah SJ, Petersson M, Maria Langkilde A, McMurray JJV, Solomon SD. Dapagliflozin and Apparent Treatment-Resistant Hypertension in Heart Failure With Mildly Reduced or Preserved Ejection Fraction: The DELIVER Trial. Circulation. 2023 Dec 12;148(24):1945-1957. doi: 10.1161/CIRCULATIONAHA.123.065254. Epub 2023 Oct 13. PMID 37830208
- [Derived] Bhatt AS, Kosiborod MN, Claggett BL, Miao ZM, Vaduganathan M, Lam CSP, Hernandez AF, Martinez FA, Inzucchi SE, Shah SJ, de Boer RA, Jhund PS, Desai AS, Fang JC, Han Y, Comin-Colet J, Drozdz J, Vardeny O, Merkely B, Lindholm D, Peterson M, Langkilde AM, McMurray JJV, Solomon SD. Impact of COVID-19 in patients with heart failure with mildly reduced or preserved ejection fraction enrolled in the DELIVER trial. Eur J Heart Fail. 2023 Dec;25(12):2177-2188. doi: 10.1002/ejhf.3043. Epub 2023 Oct 9. PMID 37771274
- [Derived] Peikert A, Bart BA, Vaduganathan M, Claggett BL, Kulac IJ, Kosiborod MN, Desai AS, Jhund PS, Lam CSP, Inzucchi SE, Martinez FA, de Boer RA, Hernandez AF, Shah SJ, Petersson M, Langkilde AM, McMurray JJV, Solomon SD, Vardeny O. Contemporary Use and Implications of Beta-Blockers in Patients With HFmrEF or HFpEF: The DELIVER Trial. JACC Heart Fail. 2024 Apr;12(4):631-644. doi: 10.1016/j.jchf.2023.09.007. Epub 2023 Sep 27. PMID 37767674
- [Derived] Chatur S, Vaduganathan M, Claggett BL, Mc Causland FR, Desai AS, Jhund PS, de Boer RA, Hernandez AF, Inzucchi SE, Kosiborod MN, Lam CSP, Martinez FA, Shah SJ, Sabatine MS, Kober L, Ponikowski P, Merkely B, Petersson M, Langkilde AM, McMurray JJV, Solomon SD. Dapagliflozin in Patients With Heart Failure and Deterioration in Renal Function. J Am Coll Cardiol. 2023 Nov 7;82(19):1854-1863. doi: 10.1016/j.jacc.2023.08.026. Epub 2023 Aug 25. PMID 37634707
- [Derived] Butt JH, Lu H, Kondo T, Bachus E, de Boer RA, Inzucchi SE, Jhund PS, Kosiborod MN, Lam CSP, Martinez FA, Vaduganathan M, Solomon SD, McMurray JJV. Heart failure, chronic obstructive pulmonary disease and efficacy and safety of dapagliflozin in heart failure with mildly reduced or preserved ejection fraction: Insights from DELIVER. Eur J Heart Fail. 2023 Nov;25(11):2078-2090. doi: 10.1002/ejhf.3000. Epub 2023 Sep 1. PMID 37634087
- [Derived] Chatur S, Vaduganathan M, Claggett BL, Cunningham JW, Docherty KF, Desai AS, Jhund PS, de Boer RA, Hernandez AF, Inzucchi SE, Kosiborod MN, Lam CSP, Martinez FA, Shah SJ, Petersson M, Langkilde AM, McMurray JJV, Solomon SD. Outpatient Worsening Among Patients With Mildly Reduced and Preserved Ejection Fraction Heart Failure in the DELIVER Trial. Circulation. 2023 Nov 28;148(22):1735-1745. doi: 10.1161/CIRCULATIONAHA.123.066506. Epub 2023 Aug 26. PMID 37632455
- [Derived] Peikert A, Goyal P, Vaduganathan M, Claggett BL, Kulac IJ, Miao ZM, Vardeny O, Kosiborod MN, Desai AS, Jhund PS, Lam CSP, Inzucchi SE, Martinez FA, de Boer RA, Hernandez AF, Shah SJ, Petersson M, Langkilde AM, McMurray JJV, Solomon SD. Dapagliflozin in Heart Failure With Mildly Reduced or Preserved Ejection Fraction According to Polypharmacy Status. JACC Heart Fail. 2023 Oct;11(10):1380-1393. doi: 10.1016/j.jchf.2023.05.014. Epub 2023 May 21. PMID 37294244
- [Derived] Ostrominski JW, Thierer J, Claggett BL, Miao ZM, Desai AS, Jhund PS, Kosiborod MN, Lam CSP, Inzucchi SE, Martinez FA, de Boer RA, Hernandez AF, Shah SJ, Petersson M, Langkilde AM, McMurray JJV, Solomon SD, Vaduganathan M. Cardio-Renal-Metabolic Overlap, Outcomes, and Dapagliflozin in Heart Failure With Mildly Reduced or Preserved Ejection Fraction. JACC Heart Fail. 2023 Nov;11(11):1491-1503. doi: 10.1016/j.jchf.2023.05.015. Epub 2023 May 24. PMID 37226448
- [Derived] Bhatt AS, Lindholm D, Nilsson A, Zaozerska N, Claggett BL, Vaduganathan M, Kosiborod MN, Lam CSP, Hernandez AF, Martinez FA, Inzucchi SE, Shah SJ, de Boer RA, Desai A, Jhund PS, Langkilde AM, Petersson M, McMurray JJV, Solomon SD. Operational challenges and mitigation measures during the COVID-19 pandemic-Lessons from DELIVER. Am Heart J. 2023 Sep;263:133-140. doi: 10.1016/j.ahj.2023.05.013. Epub 2023 May 21. PMID 37220822
- [Derived] Butt JH, Kondo T, Yang M, Jhund PS, Docherty KF, Vaduganathan M, Claggett BL, Hernandez AF, Lam CSP, Inzucchi SE, Martinez FA, de Boer RA, Kosiborod MN, Desai AS, Kober L, Ponikowski P, Sabatine MS, Shah SJ, Zaozerska N, Wilderang U, Bengtsson O, Solomon SD, McMurray JJV. Heart failure, peripheral artery disease, and dapagliflozin: a patient-level meta-analysis of DAPA-HF and DELIVER. Eur Heart J. 2023 Jun 25;44(24):2170-2183. doi: 10.1093/eurheartj/ehad276. PMID 37220172
- [Derived] Chatur S, Vaduganathan M, Claggett B, Vardeny O, Desai AS, Jhund PS, de Boer RA, Lam CSP, Kosiborod MN, Shah SJ, Martinez F, Inzucchi SE, Hernandez AF, Haddad T, Mitter SS, Miao ZM, Petersson M, Maria Langkilde A, McMurray JJV, Solomon SD. Dapagliflozin and diuretic utilization in heart failure with mildly reduced or preserved ejection fraction: the DELIVER trial. Eur Heart J. 2023 Aug 14;44(31):2930-2943. doi: 10.1093/eurheartj/ehad283. PMID 37220093
- [Derived] Chatur S, Cunningham JW, Vaduganathan M, Mc Causland FR, Claggett BL, Desai AS, Miao ZM, Jhund PS, de Boer RA, Hernandez AF, Inzucchi SE, Kosiborod MN, Lam CSP, Martinez FA, Shah SJ, Petersson M, Langkilde AM, McMurray JJV, Solomon SD. Renal and blood pressure effects of dapagliflozin in recently hospitalized patients with heart failure with mildly reduced or preserved ejection fraction: Insights from the DELIVER trial. Eur J Heart Fail. 2023 Jul;25(7):1170-1175. doi: 10.1002/ejhf.2915. Epub 2023 Jun 8. PMID 37212168
- [Derived] Bhatt AS, Kosiborod MN, Vaduganathan M, Claggett BL, Miao ZM, Kulac IJ, Lam CSP, Hernandez AF, Martinez F, Inzucchi SE, Shah SJ, de Boer RA, Jhund PS, Desai AS, Petersson M, Langkilde AM, McMurray JJV, Solomon SD. Effect of dapagliflozin on health status and quality of life across the spectrum of ejection fraction: Participant-level pooled analysis from the DAPA-HF and DELIVER trials. Eur J Heart Fail. 2023 Jul;25(7):981-988. doi: 10.1002/ejhf.2909. Epub 2023 Jun 7. PMID 37211977
- [Derived] Chatur S, Kondo T, Claggett BL, Docherty K, Miao ZM, Desai AS, Jhund PS, de Boer RA, Hernandez AF, Inzucchi SE, Kosiborod MN, Lam CSP, Martinez FA, Shah SJ, Petersson M, Langkilde AM, McMurray JJV, Solomon SD, Vaduganathan M. Effects of dapagliflozin on heart failure hospitalizations according to severity of inpatient course: Insights from DELIVER and DAPA-HF. Eur J Heart Fail. 2023 Aug;25(8):1364-1371. doi: 10.1002/ejhf.2912. Epub 2023 Jun 8. PMID 37210608
- [Derived] Peikert A, Chandra A, Kosiborod MN, Claggett BL, Desai AS, Jhund PS, Lam CSP, Inzucchi SE, Martinez FA, de Boer RA, Hernandez AF, Shah SJ, Janssens SP, Belohlavek J, Borleffs CJW, Dobreanu D, Langkilde AM, Bengtsson O, Petersson M, McMurray JJV, Solomon SD, Vaduganathan M. Association of Dapagliflozin vs Placebo With Individual Kansas City Cardiomyopathy Questionnaire Components in Patients With Heart Failure With Mildly Reduced or Preserved Ejection Fraction: A Secondary Analysis of the DELIVER Trial. JAMA Cardiol. 2023 Jul 1;8(7):684-690. doi: 10.1001/jamacardio.2023.1342. PMID 37208998
- [Derived] Jhund PS, Claggett BL, Talebi A, Butt JH, Gasparyan SB, Wei LJ, McCaw ZR, Wilderang U, Bengtsson O, Desai AS, Petersson M, Langkilde AM, de Boer RA, Hernandez AF, Inzucchi SE, Kosiborod MN, Lam CSP, Martinez FA, Shah SJ, Vaduganathan M, Solomon SD, McMurray JJV. Effect of Dapagliflozin on Total Heart Failure Events in Patients With Heart Failure With Mildly Reduced or Preserved Ejection Fraction: A Prespecified Analysis of the DELIVER Trial. JAMA Cardiol. 2023 Jun 1;8(6):554-563. doi: 10.1001/jamacardio.2023.0711. PMID 37099283
- [Derived] Vaduganathan M, Claggett BL, Jhund P, Miao ZM, de Boer RA, Lam CSP, Desai AS, Bengsston O, McMurray JJV, Solomon SD. Dapagliflozin and All-Cause Hospitalizations in Patients With Heart Failure With Preserved Ejection Fraction. J Am Coll Cardiol. 2023 Mar 14;81(10):1004-1006. doi: 10.1016/j.jacc.2022.12.026. No abstract available. PMID 36889870
- [Derived] Butt JH, Docherty KF, Claggett BL, Desai AS, Fang JC, Petersson M, Langkilde AM, de Boer RA, Cabrera Honorio JW, Hernandez AF, Inzucchi SE, Kosiborod MN, Kober L, Lam CSP, Martinez FA, Ponikowski P, Sabatine MS, Vardeny O, O'Meara E, Saraiva JFK, Shah SJ, Vaduganathan M, Jhund PS, Solomon SD, McMurray JJV. Dapagliflozin in Black and White Patients With Heart Failure Across the Ejection Fraction Spectrum. JACC Heart Fail. 2023 Apr;11(4):375-388. doi: 10.1016/j.jchf.2022.11.014. Epub 2023 Feb 1. PMID 36881399
- [Derived] Kondo T, Jering KS, Borleffs CJW, de Boer RA, Claggett BL, Desai AS, Dobreanu D, Inzucchi SE, Hernandez AF, Janssens SP, Jhund PS, Kosiborod MN, Lam CSP, Langkilde AM, Martinez FA, Petersson M, Vinh PN, Vaduganathan M, Solomon SD, McMurray JJV. Patient Characteristics, Outcomes, and Effects of Dapagliflozin According to the Duration of Heart Failure: A Prespecified Analysis of the DELIVER Trial. Circulation. 2023 Apr 4;147(14):1067-1078. doi: 10.1161/CIRCULATIONAHA.122.062918. Epub 2023 Mar 6. PMID 36876483
- [Derived] Butt JH, Docherty KF, Claggett BL, Desai AS, Petersson M, Langkilde AM, de Boer RA, Hernandez AF, Inzucchi SE, Kosiborod MN, Kober L, Lam CSP, Martinez FA, Ponikowski P, Sabatine MS, Shah SJ, Vaduganathan M, Jhund PS, Solomon SD, McMurray JJV. Association of Dapagliflozin Use With Clinical Outcomes and the Introduction of Uric Acid-Lowering Therapy and Colchicine in Patients With Heart Failure With and Without Gout: A Patient-Level Pooled Meta-analysis of DAPA-HF and DELIVER. JAMA Cardiol. 2023 Apr 1;8(4):386-393. doi: 10.1001/jamacardio.2022.5608. PMID 36811901
- [Derived] Selvaraj S, Vaduganathan M, Claggett BL, Miao ZM, Fang JC, Vardeny O, Desai AS, Shah SJ, Lam CSP, Martinez FA, Inzucchi SE, de Boer RA, Petersson M, Langkilde AM, McMurray JJV, Solomon SD. Blood Pressure and Dapagliflozin in Heart Failure With Mildly Reduced or Preserved Ejection Fraction: DELIVER. JACC Heart Fail. 2023 Jan;11(1):76-89. doi: 10.1016/j.jchf.2022.09.002. Epub 2022 Oct 2. PMID 36599553
- [Derived] Kosiborod MN, Bhatt AS, Claggett BL, Vaduganathan M, Kulac IJ, Lam CSP, Hernandez AF, Martinez FA, Inzucchi SE, Shah SJ, de Boer RA, Jhund PS, Desai AS, Fang JC, Han Y, Comin-Colet J, Vardeny O, Lindholm D, Wilderang U, Bengtsson O, McMurray JJV, Solomon SD. Effect of Dapagliflozin on Health Status in Patients With Preserved or Mildly Reduced Ejection Fraction. J Am Coll Cardiol. 2023 Feb 7;81(5):460-473. doi: 10.1016/j.jacc.2022.11.006. Epub 2022 Dec 14. PMID 36526515
- [Derived] Vardeny O, Fang JC, Desai AS, Jhund PS, Claggett B, Vaduganathan M, de Boer RA, Hernandez AF, Lam CSP, Inzucchi SE, Martinez FA, Kosiborod MN, DeMets D, O'Meara E, Zieroth S, Comin-Colet J, Drozdz J, Chiang CE, Kitakaze M, Petersson M, Lindholm D, Langkilde AM, McMurray JJV, Solomon SD. Dapagliflozin in heart failure with improved ejection fraction: a prespecified analysis of the DELIVER trial. Nat Med. 2022 Dec;28(12):2504-2511. doi: 10.1038/s41591-022-02102-9. Epub 2022 Dec 15. PMID 36522606
- [Derived] Inzucchi SE, Claggett BL, Vaduganathan M, Desai AS, Jhund PS, de Boer RA, Hernandez AF, Kosiborod MN, Lam CSP, Martinez F, Shah SJ, Verma S, Han Y, Kerr Saraiva JF, Bengtsson O, Petersson M, Langkilde AM, McMurray JJV, Solomon SD. Efficacy and safety of dapagliflozin in patients with heart failure with mildly reduced or preserved ejection fraction by baseline glycaemic status (DELIVER): a subgroup analysis from an international, multicentre, double-blind, randomised, placebo-controlled trial. Lancet Diabetes Endocrinol. 2022 Dec;10(12):869-881. doi: 10.1016/S2213-8587(22)00308-4. Epub 2022 Nov 10. PMID 36372069
- [Derived] Mc Causland FR, Claggett BL, Vaduganathan M, Desai AS, Jhund P, de Boer RA, Docherty K, Fang J, Hernandez AF, Inzucchi SE, Kosiborod MN, Lam CSP, Martinez F, Saraiva JFK, McGrath MM, Shah SJ, Verma S, Langkilde AM, Petersson M, McMurray JJV, Solomon SD. Dapagliflozin and Kidney Outcomes in Patients With Heart Failure With Mildly Reduced or Preserved Ejection Fraction: A Prespecified Analysis of the DELIVER Randomized Clinical Trial. JAMA Cardiol. 2023 Jan 1;8(1):56-65. doi: 10.1001/jamacardio.2022.4210. PMID 36326604
- [Derived] Vaduganathan M, Claggett BL, Jhund P, de Boer RA, Hernandez AF, Inzucchi SE, Kosiborod MN, Lam CSP, Martinez F, Shah SJ, Desai AS, Hegde SM, Lindholm D, Petersson M, Langkilde AM, McMurray JJV, Solomon SD. Time to Clinical Benefit of Dapagliflozin in Patients With Heart Failure With Mildly Reduced or Preserved Ejection Fraction: A Prespecified Secondary Analysis of the DELIVER Randomized Clinical Trial. JAMA Cardiol. 2022 Dec 1;7(12):1259-1263. doi: 10.1001/jamacardio.2022.3750. PMID 36190011
- [Derived] Desai AS, Jhund PS, Claggett BL, Vaduganathan M, Miao ZM, Kondo T, Barkoudah E, Brahimi A, Connolly E, Finn P, Lang NN, Mc Causland FR, McGrath M, Petrie MC, McMurray JJV, Solomon SD. Effect of Dapagliflozin on Cause-Specific Mortality in Patients With Heart Failure Across the Spectrum of Ejection Fraction: A Participant-Level Pooled Analysis of DAPA-HF and DELIVER. JAMA Cardiol. 2022 Dec 1;7(12):1227-1234. doi: 10.1001/jamacardio.2022.3736. PMID 36189985
- [Derived] Myhre PL, Vaduganathan M, Claggett BL, Miao ZM, Jhund PS, de Boer RA, Hernandez AF, Inzucchi SE, Kosiborod MN, Lam CSP, Martinez F, Shah SJ, Desai AS, Lindholm D, Petersson M, Langkilde AM, McMurray JJV, Solomon SD. Influence of NT-proBNP on Efficacy of Dapagliflozin in Heart Failure With Mildly Reduced or Preserved Ejection Fraction. JACC Heart Fail. 2022 Dec;10(12):902-913. doi: 10.1016/j.jchf.2022.08.007. Epub 2022 Aug 27. PMID 36114137
- [Derived] Peters AE, Ogunniyi MO, Hegde SM, Bianco C, Ghafghazi S, Hernandez AF, DeVore AD. A multicenter program for electronic health record screening for patients with heart failure with preserved ejection fraction: Lessons from the DELIVER-EHR initiative. Contemp Clin Trials. 2022 Oct;121:106924. doi: 10.1016/j.cct.2022.106924. Epub 2022 Sep 12. PMID 36100197
- [Derived] Cunningham JW, Vaduganathan M, Claggett BL, Kulac IJ, Desai AS, Jhund PS, de Boer RA, DeMets D, Hernandez AF, Inzucchi SE, Kosiborod MN, Lam CSP, Martinez F, Shah SJ, McGrath MM, O'Meara E, Wilderang U, Lindholm D, Petersson M, Langkilde AM, McMurray JJV, Solomon SD. Dapagliflozin in Patients Recently Hospitalized With Heart Failure and Mildly Reduced or Preserved Ejection Fraction. J Am Coll Cardiol. 2022 Oct 4;80(14):1302-1310. doi: 10.1016/j.jacc.2022.07.021. Epub 2022 Aug 27. PMID 36041912
- [Derived] Vaduganathan M, Claggett BL, Jhund P, de Boer RA, Hernandez AF, Inzucchi SE, Kosiborod MN, Lam CSP, Martinez F, Shah SJ, Desai AS, Lindholm D, Petersson M, Langkilde AM, McMurray JJV, Solomon SD. Estimated Long-Term Benefit of Dapagliflozin in Patients With Heart Failure. J Am Coll Cardiol. 2022 Nov 8;80(19):1775-1784. doi: 10.1016/j.jacc.2022.08.745. Epub 2022 Aug 27. PMID 36041669
- [Derived] Butt JH, Kondo T, Jhund PS, Comin-Colet J, de Boer RA, Desai AS, Hernandez AF, Inzucchi SE, Janssens SP, Kosiborod MN, Lam CSP, Langkilde AM, Lindholm D, Martinez F, Petersson M, Shah SJ, Thierer J, Vaduganathan M, Verma S, Wilderang U, Claggett BC, Solomon SD, McMurray JJV. Atrial Fibrillation and Dapagliflozin Efficacy in Patients With Preserved or Mildly Reduced Ejection Fraction. J Am Coll Cardiol. 2022 Nov 1;80(18):1705-1717. doi: 10.1016/j.jacc.2022.08.718. Epub 2022 Aug 27. PMID 36041668
- [Derived] Peikert A, Martinez FA, Vaduganathan M, Claggett BL, Kulac IJ, Desai AS, Jhund PS, de Boer RA, DeMets D, Hernandez AF, Inzucchi SE, Kosiborod MN, Lam CSP, Shah SJ, Katova T, Merkely B, Vardeny O, Wilderang U, Lindholm D, Petersson M, Langkilde AM, McMurray JJV, Solomon SD. Efficacy and Safety of Dapagliflozin in Heart Failure With Mildly Reduced or Preserved Ejection Fraction According to Age: The DELIVER Trial. Circ Heart Fail. 2022 Oct;15(10):e010080. doi: 10.1161/CIRCHEARTFAILURE.122.010080. Epub 2022 Aug 27. PMID 36029467
- [Derived] Butt JH, Jhund PS, Belohlavek J, de Boer RA, Chiang CE, Desai AS, Drozdz J, Hernandez AF, Inzucchi SE, Katova T, Kitakaze M, Kosiborod MN, Lam CSP, Maria Langkilde A, Lindholm D, Bachus E, Martinez F, Merkely B, Petersson M, Saraiva JFK, Shah SJ, Vaduganathan M, Vardeny O, Wilderang U, Claggett BL, Solomon SD, McMurray JJV. Efficacy and Safety of Dapagliflozin According to Frailty in Patients With Heart Failure: A Prespecified Analysis of the DELIVER Trial. Circulation. 2022 Oct 18;146(16):1210-1224. doi: 10.1161/CIRCULATIONAHA.122.061754. Epub 2022 Aug 27. PMID 36029465
- [Derived] Solomon SD, McMurray JJV, Claggett B, de Boer RA, DeMets D, Hernandez AF, Inzucchi SE, Kosiborod MN, Lam CSP, Martinez F, Shah SJ, Desai AS, Jhund PS, Belohlavek J, Chiang CE, Borleffs CJW, Comin-Colet J, Dobreanu D, Drozdz J, Fang JC, Alcocer-Gamba MA, Al Habeeb W, Han Y, Cabrera Honorio JW, Janssens SP, Katova T, Kitakaze M, Merkely B, O'Meara E, Saraiva JFK, Tereshchenko SN, Thierer J, Vaduganathan M, Vardeny O, Verma S, Pham VN, Wilderang U, Zaozerska N, Bachus E, Lindholm D, Petersson M, Langkilde AM; DELIVER Trial Committees and Investigators. Dapagliflozin in Heart Failure with Mildly Reduced or Preserved Ejection Fraction. N Engl J Med. 2022 Sep 22;387(12):1089-1098. doi: 10.1056/NEJMoa2206286. Epub 2022 Aug 27. PMID 36027570
- [Derived] Solomon SD, Vaduganathan M, Claggett BL, de Boer RA, DeMets D, Hernandez AF, Inzucchi SE, Kosiborod MN, Lam CSP, Martinez F, Shah SJ, Belohlavek J, Chiang CE, Willem Borleffs CJ, Comin-Colet J, Dobreanu D, Drozdz J, Fang JC, Alcocer Gamba MA, Al Habeeb W, Han Y, Cabrera Honorio JW, Janssens SP, Katova T, Kitakaze M, Merkely B, O'Meara E, Kerr Saraiva JF, Tereschenko SN, Thierer J, Vardeny O, Verma S, Vinh PN, Wilderang U, Zaozerska N, Lindholm D, Petersson M, McMurray JJV. Baseline Characteristics of Patients With HF With Mildly Reduced and Preserved Ejection Fraction: DELIVER Trial. JACC Heart Fail. 2022 Mar;10(3):184-197. doi: 10.1016/j.jchf.2021.11.006. PMID 35241246
- [Derived] Kanie T, Mizuno A, Takaoka Y, Suzuki T, Yoneoka D, Nishikawa Y, Tam WWS, Morze J, Rynkiewicz A, Xin Y, Wu O, Providencia R, Kwong JS. Dipeptidyl peptidase-4 inhibitors, glucagon-like peptide 1 receptor agonists and sodium-glucose co-transporter-2 inhibitors for people with cardiovascular disease: a network meta-analysis. Cochrane Database Syst Rev. 2021 Oct 25;10(10):CD013650. doi: 10.1002/14651858.CD013650.pub2. PMID 34693515
- [Derived] Nassif ME, Kosiborod M. Effects of sodium glucose cotransporter type 2 inhibitors on heart failure. Diabetes Obes Metab. 2019 Apr;21 Suppl 2:19-23. doi: 10.1111/dom.13678. PMID 31081589
- See also: Redacted Clinical Study Protocol — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D169CC00001&attachmentIdentifier=219ed7c1-2b33-4f6b-be14-6261816c74e8&fileName=D169CC00001_DELIVER_CSP_12Nov2020_version_4.0_Redacted2.pdf&versionIdentifier=
- See also: Redacted Statistical Analysis Plan — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D169CC00001&attachmentIdentifier=8cd4f2a7-521d-4001-9dfc-351e1b077a4d&fileName=D169CC00001_-___Statistical_Analysis_Plan_v5.0_Redacted.pdf&versionIdentifier=
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D169CC00001&attachmentIdentifier=6d2e647c-a9ac-445e-b0b8-91a252dcd8a4&fileName=D169CC00001-CSR-Synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Dapa 10 mg: Dapagliflozin 10 mg tablets administered once daily per oral use
- Placebo: Placebo tablet to match dapagliflozin 10 mg, given once daily per oral use
Period: Overall Study
Arm/Group | Dapa 10 mg | Placebo
Started | 3131 | 3132
Completed | 3121 | 3121
Not Completed | 10 | 11
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 8 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapa 10 mg | Placebo | Total
Number analyzed (Participants) | 3131 | 3132 | 6263
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.8 (9.6) | 71.5 (9.5) | 71.7 (9.6)
Age, Customized [Count of Participants; unit: Participants]
  <= 50 | 85 | 74 | 159
  > 50 | 3046 | 3058 | 6104
Age, Customized [Count of Participants; unit: Participants]
  <= 65 | 743 | 761 | 1504
  > 65 | 2388 | 2371 | 4759
Age, Customized [Count of Participants; unit: Participants]
  <= 65 | 743 | 761 | 1504
  >65 - 75 | 1184 | 1228 | 2412
  > 75 | 1204 | 1143 | 2347
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1364 | 1383 | 2747
  Male | 1767 | 1749 | 3516
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 632 | 598 | 1230
  Not Hispanic or Latino | 2499 | 2534 | 5033
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2214 | 2225 | 4439
  Black or African American | 81 | 78 | 159
  Asian | 630 | 644 | 1274
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0
  American Indian or Alaska Native | 93 | 96 | 189
  Other | 113 | 89 | 202
Prior HF Hospitalization [Count of Participants; unit: Participants]
  Yes | 1270 | 1269 | 2539
NYHA Class at Baseline [Count of Participants; unit: Participants] — NYHA functional classification: I No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnoea (shortness of breath). II Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea. III Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea. IV Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases.
  Participants
    I | 0 | 1 | 1
    II | 2314 | 2399 | 4713
    III | 807 | 724 | 1531
    IV | 10 | 8 | 18
Medical History of Type 2 Diabetes [Count of Participants; unit: Participants]
  Yes | 1401 | 1405 | 2806
LVEF (%) at Baseline [Mean (Standard Deviation); unit: Percentage of blood leaving the heart] | 54.0 (8.6) | 54.3 (8.9) | 54.2 (8.8)

OUTCOME MEASURES:

1. Primary Outcome: Subjects Included in the Composite Endpoint of CV Death, Hospitalization Due to Heart Failure or Urgent Visit Due to Heart Failure.
Description: Dual primary efficacy
  Primary endpoint analysed in all patients randomised (Full analysis set).
  The analysis was assessed on Full Analysis Set, including events occurring on or prior to Primary Analysis Censoring Date.
Time Frame: Up to 42.1 months
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Dapa 10 mg | Placebo
Number analyzed (Participants) | 3131 | 3132
Participants | 512 | 610
Statistical Analysis 1: Comparison: Dapa 10 mg vs Placebo; Comparison Group: Placebo; Test type: Superiority; p = 0.0008, Regression, Cox; Stratified by Type 2 Diabetes status at randomization; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.73 to 0.92]

2. Primary Outcome: Subjects Included in the Composite Endpoint of CV Death, Hospitalization Due to Heart Failure or Urgent Visit Due to Heart Failure for LVEF <60% Subpopulation
Description: Dual primary efficacy
  Primary endpoint analysed in all patients randomised with LVEF < 60% at baseline.
  The analysis was assessed on Full Analysis Set, including events occurring on or prior to Primary Analysis Censoring Date.
Time Frame: Up to 42.1 months
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Dapa 10 mg | Placebo
Number analyzed (Participants) | 2200 | 2172
Participants | 381 | 440
Statistical Analysis 1: Comparison: Dapa 10 mg vs Placebo; Comparison Group: Placebo; Test type: Superiority; p = 0.0085, Regression, Cox; Stratified by Type 2 Diabetes status at randomization; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.73 to 0.95]

3. Secondary Outcome: Events Included in the Composite Endpoint of CV Death or Recurrent Heart Failure Event (Hospitalization Due to Heart Failure or Urgent Heart Failure Visit)
Description: Secondary efficacy
  Total number of heart failure events (first and recurrent) and cardiovascular death, analysed in all randomized patients.
  The analysis was assessed on Full Analysis Set, including events occurring on or prior to Primary Analysis Censoring Date.
Time Frame: Up to 42.1 months
Population: Full analysis set population
Measure: Number; unit: Number of events
Arm/Group | Dapa 10 mg | Placebo
Number analyzed (Participants) | 3131 | 3132
Number of events | 815 | 1057
Statistical Analysis 1: Comparison: Dapa 10 mg vs Placebo; Comparison Group: Placebo; Test type: Superiority; p = 0.0003, LWYY proportional rates model; Stratified by Type 2 Diabetes status at randomization; Rate Ratio (RR) = 0.77, 95% CI 2-sided [0.67 to 0.89]

4. Secondary Outcome: Events Included in the Composite Endpoint of CV Death or Recurrent Heart Failure Event (Hospitalization Due to Heart Failure or Urgent Heart Failure Visit) for LVEF <60% Subpopulation
Description: Secondary efficacy
  Total number of heart failure events (first and recurrent) and cardiovascular death, analysed in all randomized patients with LVEF < 60% at baseline
  The analysis was assessed on Full Analysis Set, including events occurring on or prior to Primary Analysis Censoring Date.
Time Frame: Up to 42.1 months
Population: Full analysis set population
Measure: Number; unit: Number of events
Arm/Group | Dapa 10 mg | Placebo
Number analyzed (Participants) | 2200 | 2172
Number of events | 605 | 782
Statistical Analysis 1: Comparison: Dapa 10 mg vs Placebo; Comparison Group: Placebo; Test type: Superiority; p = 0.0017, LWYY proportional rates model; Stratified by Type 2 Diabetes status at randomization; Rate Ratio (RR) = 0.77, 95% CI 2-sided [0.65 to 0.90]

5. Secondary Outcome: Change From Baseline in the KCCQ Total Symptom Score at 8 Months
Description: KCCQ is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. The KCCQ Total Symptom Score incorporates the symptom domains into a single score. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Time Frame: Baseline and 8 months or death before 8 months
Population: Full analysis set population, including only assessments performed or planned prior to March 11th, 2020, when COVID-19 was declared a pandemic by the WHO.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Dapa 10 mg | Placebo
Number analyzed (Participants) | 1316 | 1311
Scores on a scale | 8.3 (20.3) | 5.2 (21.1)
Statistical Analysis 1: Comparison: Dapa 10 mg vs Placebo; Comparison Group: Placebo; Test type: Superiority; p = 0.0086, Win Ratio — The p-value is obtained from a rank ANCOVA adjusted for baseline KCCQ score, stratified by T2DM status at randomisation; Stratified by Type 2 Diabetes status at randomization and including baseline score as a covariate; Rate Ratio (RR) = 1.11, 95% CI 2-sided [1.03 to 1.21] — The composite of change from baseline in KCCQ Total Symptom Score at 8 months, or death before 8 months

6. Secondary Outcome: Subjects Included in the Endpoint of Cardiovascular Death
Description: Secondary efficacy
  The analysis was assessed on Full Analysis Set, including deaths occurring on or prior to Primary Analysis Censoring Date.
Time Frame: Up to 42.1 months
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Dapa 10 mg | Placebo
Number analyzed (Participants) | 3131 | 3132
Participants | 231 | 261
Statistical Analysis 1: Comparison: Dapa 10 mg vs Placebo; Comparison Group: Placebo; Test type: Superiority; p = 0.1678, Regression, Cox; Stratified by Type 2 Diabetes status at randomization; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.74 to 1.05]

7. Secondary Outcome: Subjects Included in the Endpoint of All-cause Mortality
Description: as for outcome 6
Time Frame: Up to 42.1 months
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Dapa 10 mg | Placebo
Number analyzed (Participants) | 3131 | 3132
Participants | 497 | 526
Statistical Analysis 1: Comparison: Dapa 10 mg vs Placebo; Comparison Group: Placebo; Test type: Superiority; p = 0.3425, Regression, Cox; Stratified by Type 2 Diabetes status at randomization; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.83 to 1.07]

ADVERSE EVENTS:
Time Frame: [All-cause mortality]: From randomization until end of study, up to 42.2 months. [Serious AE and other AE] From first dose until end of study, up to 42.2 months.
Description: [All-cause mortality]: Full analysis set (all randomized patients). [Serious AE and other AE] Safety analysis set (patients who received at least 1 dose of study drug).
  Serious AEs, AEs leading to discontinuation/ amputation/ preceding events/ potential endpoint/ interruption of study drug, non-serious AEs including myocardial infarction, unstable angina, stroke, major hypoglycaemic events, potential DKA and amputation were collected systematically. Other AEs were non-systematically collected.
Arm/Group | Dapa 10 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 510/3131 | 533/3132
Serious Adverse Events (participants affected / at risk) | 1454/3126 | 1508/3127
Other Adverse Events (participants affected / at risk) | 464/3126 | 485/3127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapa 10 mg (N=3126) | Placebo (N=3127)
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (3) | 3 (3)
Vertigo positional (Ear and labyrinth disorders) | 3 (3) | 1 (1)
Goitre (Endocrine disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 2 (2)
Age-related macular degeneration (Eye disorders) | 0 (0) | 1 (1)
Amaurosis fugax (Eye disorders) | 1 (1) | 0 (0)
Hypocoagulable state (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Blindness (Eye disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 10 (12) | 5 (7)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 2 (2) | 0 (0)
Epiretinal membrane (Eye disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 1 (1)
Lens dislocation (Eye disorders) | 1 (1) | 0 (0)
Macular rupture (Eye disorders) | 0 (0) | 1 (2)
Retinal artery occlusion (Eye disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 2 (2) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3 (3) | 5 (5)
Visual impairment (Eye disorders) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 2 (2)
Vitreous opacities (Eye disorders) | 1 (1) | 0 (0)
Abdominal adhesions (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal incarcerated hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 4 (4)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute abdomen (Gastrointestinal disorders) | 0 (0) | 2 (2)
Anal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 4 (5)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (1) | 8 (8)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 2 (2)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 4 (4)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 2 (2) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 2 (2)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (2)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterovesical fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Erosive duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric antral vascular ectasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastric ulcer (Gastrointestinal disorders) | 3 (3) | 5 (5)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 2 (2) | 3 (3)
Gastritis (Gastrointestinal disorders) | 3 (4) | 2 (2)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (2)
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 2 (2)
Normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 14 (14) | 15 (17)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal vascular malformation haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 3 (3)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (2) | 1 (1)
Haemoperitoneum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 3 (3)
Ileal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 3 (3)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 6 (7) | 5 (5)
Inguinal hernia strangulated (Gastrointestinal disorders) | 1 (1) | 0 (0)
Splenic cyst (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Intestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 3 (3)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 5 (5)
Intra-abdominal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ischaemic enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 11 (12)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 (5) | 4 (5)
Mechanical ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (2) | 2 (2)
Mesenteric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Obstructive pancreatitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Oesophageal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatic duct dilatation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 3 (3)
Pancreatitis acute (Gastrointestinal disorders) | 2 (2) | 7 (8)
Anaemia (Blood and lymphatic system disorders) | 16 (18) | 24 (26)
Acute coronary syndrome (Cardiac disorders) | 2 (2) | 1 (1)
Pancreatitis chronic (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pancreatitis necrotising (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Rectal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 1 (1)
Salivary gland calculus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (4) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 10 (12) | 16 (19)
Strangulated umbilical hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Stress ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tooth impacted (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical hernia, obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (4) | 7 (7)
Volvulus (Gastrointestinal disorders) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Asthenia (General disorders) | 5 (5) | 4 (4)
Acute myocardial infarction (Cardiac disorders) | 63 (73) | 63 (71)
Cardiac death (General disorders) | 3 (3) | 3 (3)
Catheter site pain (General disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 7 (8) | 9 (9)
Death (General disorders) | 54 (54) | 52 (52)
Feeling abnormal (General disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 1 (1)
Hypothermia (General disorders) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 1 (1) | 0 (0)
Acute right ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Incarcerated hernia (General disorders) | 1 (1) | 0 (0)
Inflammation (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 2 (2)
Medical device site joint inflammation (General disorders) | 1 (1) | 0 (0)
Multimorbidity (General disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 3 (3) | 3 (3)
Non-cardiac chest pain (General disorders) | 7 (11) | 7 (8)
Oedema due to cardiac disease (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 18 (20) | 19 (21)
Procedural failure (General disorders) | 1 (1) | 0 (0)
Prosthetic cardiac valve thrombosis (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 2 (2)
Stent-graft endoleak (General disorders) | 1 (1) | 0 (0)
Sudden cardiac death (General disorders) | 26 (26) | 37 (37)
Sudden death (General disorders) | 24 (24) | 26 (26)
Ulcer haemorrhage (General disorders) | 1 (1) | 0 (0)
Vascular stent stenosis (General disorders) | 1 (1) | 0 (0)
Vascular stent thrombosis (General disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 4 (5) | 1 (1)
Angina unstable (Cardiac disorders) | 49 (56) | 62 (75)
Biliary colic (Hepatobiliary disorders) | 1 (2) | 0 (0)
Biliary dilatation (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 2 (2) | 3 (3)
Cholangitis acute (Hepatobiliary disorders) | 2 (4) | 3 (3)
Cholecystitis (Hepatobiliary disorders) | 8 (8) | 7 (8)
Cholecystitis acute (Hepatobiliary disorders) | 3 (3) | 6 (6)
Cholecystitis chronic (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 5 (5) | 3 (3)
Congestive hepatopathy (Hepatobiliary disorders) | 2 (2) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 2 (2) | 4 (4)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatic mass (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis alcoholic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 2 (2) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Amyloidosis (Immune system disorders) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 6 (6)
Contrast media allergy (Immune system disorders) | 2 (2) | 0 (0)
Heart transplant rejection (Immune system disorders) | 0 (0) | 1 (1)
Primary amyloidosis (Immune system disorders) | 1 (1) | 0 (0)
Abdominal sepsis (Infections and infestations) | 1 (1) | 1 (1)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 2 (3)
Acinetobacter sepsis (Infections and infestations) | 0 (0) | 1 (1)
Acute endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 6 (6)
Arrhythmia (Cardiac disorders) | 1 (1) | 2 (2)
Appendicitis perforated (Infections and infestations) | 1 (1) | 3 (3)
Arthritis bacterial (Infections and infestations) | 1 (1) | 1 (1)
Asymptomatic covid-19 (Infections and infestations) | 24 (25) | 23 (23)
Atypical pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Bacteraemia (Infections and infestations) | 2 (2) | 1 (1)
Bacterial prostatitis (Infections and infestations) | 1 (1) | 0 (0)
Bacterial pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Biliary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 8 (8) | 12 (14)
Bronchitis viral (Infections and infestations) | 2 (2) | 0 (0)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1) | 0 (0)
Bullous erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Bursitis infective (Infections and infestations) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 183 (187) | 144 (147)
Covid-19 pneumonia (Infections and infestations) | 86 (86) | 89 (91)
Cellulitis (Infections and infestations) | 35 (44) | 22 (30)
Cholangitis infective (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 2 (2) | 2 (2)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 4 (4)
Complicated appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Coronavirus infection (Infections and infestations) | 0 (0) | 2 (2)
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 69 (82) | 57 (62)
Coronavirus pneumonia (Infections and infestations) | 3 (3) | 2 (2)
Cystitis (Infections and infestations) | 3 (3) | 2 (2)
Cystitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Cystitis escherichia (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 2 (2) | 0 (0)
Device related sepsis (Infections and infestations) | 0 (0) | 1 (1)
Diabetic foot infection (Infections and infestations) | 2 (2) | 2 (4)
Diabetic gangrene (Infections and infestations) | 1 (1) | 2 (4)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 4 (4) | 5 (5)
Atrial flutter (Cardiac disorders) | 10 (10) | 2 (2)
Diverticulitis intestinal perforated (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 2 (2) | 3 (3)
Endocarditis bacterial (Infections and infestations) | 1 (1) | 1 (1)
Endocarditis enterococcal (Infections and infestations) | 0 (0) | 2 (2)
Enterococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 6 (6) | 4 (4)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 2 (2)
Escherichia sepsis (Infections and infestations) | 1 (1) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 6 (7) | 1 (1)
Furuncle (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 4 (4) | 4 (4)
Gastroenteritis (Infections and infestations) | 7 (7) | 8 (8)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 2 (2)
Hiv infection (Infections and infestations) | 0 (0) | 1 (1)
Haematoma infection (Infections and infestations) | 1 (1) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis c (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis e (Infections and infestations) | 0 (0) | 1 (1)
Atrial thrombosis (Cardiac disorders) | 2 (2) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 2 (2)
Herpes zoster disseminated (Infections and infestations) | 1 (1) | 0 (0)
Implant site infection (Infections and infestations) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 1 (1) | 4 (4)
Infection (Infections and infestations) | 1 (1) | 3 (3)
Infectious pleural effusion (Infections and infestations) | 3 (3) | 2 (2)
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 4 (4) | 5 (5)
Intestinal gangrene (Infections and infestations) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 1 (1) | 3 (3)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 1 (1)
Large intestine infection (Infections and infestations) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 2 (2) | 0 (0)
Localised infection (Infections and infestations) | 3 (3) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 3 (4)
Lower respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Lung abscess (Infections and infestations) | 1 (1) | 1 (1)
Lymph node tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Mediastinitis (Infections and infestations) | 0 (0) | 1 (1)
Middle east respiratory syndrome (Infections and infestations) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 7 (7) | 4 (4)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 1 (1)
Ophthalmic herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 7 (7) | 7 (8)
Osteomyelitis chronic (Infections and infestations) | 1 (1) | 0 (0)
Pancreas infection (Infections and infestations) | 0 (0) | 1 (1)
Pelvic abscess (Infections and infestations) | 0 (0) | 1 (1)
Pelvic inflammatory disease (Infections and infestations) | 0 (0) | 1 (1)
Periodontitis (Infections and infestations) | 1 (1) | 2 (2)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 1 (1)
Peritonitis (Infections and infestations) | 2 (2) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Peritonsillar abscess (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 113 (123) | 106 (129)
Pneumonia aspiration (Infections and infestations) | 7 (7) | 8 (8)
Pneumonia bacterial (Infections and infestations) | 3 (3) | 7 (7)
Pneumonia pseudomonal (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 3 (3)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Atrioventricular dissociation (Cardiac disorders) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 3 (3) | 1 (1)
Prosthetic valve endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 2 (2) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 2 (2) | 3 (4)
Pyelonephritis acute (Infections and infestations) | 2 (2) | 0 (0)
Pyelonephritis chronic (Infections and infestations) | 2 (2) | 0 (0)
Respiratory syncytial virus bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 4 (4)
Sepsis (Infections and infestations) | 16 (17) | 20 (21)
Bradyarrhythmia (Cardiac disorders) | 2 (2) | 2 (2)
Septic phlebitis (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 17 (17) | 17 (18)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 2 (2) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Spontaneous bacterial peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Staphylococcal infection (Infections and infestations) | 2 (2) | 2 (2)
Streptococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 11 (11) | 13 (13)
Suspected covid-19 (Infections and infestations) | 17 (17) | 16 (16)
Testicular abscess (Infections and infestations) | 0 (0) | 1 (1)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1)
Tuberculosis (Infections and infestations) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 2 (2)
Urinary tract infection (Infections and infestations) | 40 (49) | 33 (34)
Urosepsis (Infections and infestations) | 8 (8) | 11 (12)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Viral myositis (Infections and infestations) | 1 (1) | 0 (0)
Viral pericarditis (Infections and infestations) | 1 (1) | 0 (0)
Blood loss anaemia (Blood and lymphatic system disorders) | 4 (4) | 6 (6)
Bundle branch block left (Cardiac disorders) | 0 (0) | 2 (2)
Vulval cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 2 (2) | 3 (3)
Wound sepsis (Infections and infestations) | 0 (0) | 1 (1)
Abdominal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Brain contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cardiac amyloidosis (Cardiac disorders) | 0 (0) | 1 (1)
Burns third degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Comminuted fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Compression fracture (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Coronary bypass stenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 18 (18) | 17 (17)
Eschar (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 5 (5) | 7 (7)
Femoral neck fracture (Injury, poisoning and procedural complications) | 6 (6) | 5 (5)
Femur fracture (Injury, poisoning and procedural complications) | 10 (10) | 11 (12)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fractured sacrum (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Cardiac disorder (Cardiac disorders) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 6 (6)
Heat illness (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 10 (10) | 7 (7)
Humerus fracture (Injury, poisoning and procedural complications) | 3 (3) | 6 (6)
Incarcerated incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 308 (458) | 377 (581)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Open fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Penis injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 57 (73) | 63 (90)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post procedural hypotension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural swelling (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Repetitive strain injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 23 (32) | 26 (44)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Road traffic accident (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 11 (11) | 5 (5)
Spinal cord injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Splenic rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stomal hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 4 (4) | 4 (4)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 63 (86) | 82 (116)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (4)
Vascular graft stenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Cardiac failure high output (Cardiac disorders) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anticoagulation drug level above therapeutic (Investigations) | 0 (0) | 2 (2)
Blood creatinine increased (Investigations) | 1 (2) | 0 (0)
Ejection fraction decreased (Investigations) | 2 (2) | 1 (1)
Electrocardiogram qrs complex prolonged (Investigations) | 1 (1) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 1 (1) | 0 (0)
Fibrin d dimer increased (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1)
Cardiac valve disease (Cardiac disorders) | 2 (2) | 3 (3)
Peripheral pulse decreased (Investigations) | 1 (1) | 0 (0)
Sars-cov-2 antibody test positive (Investigations) | 0 (0) | 1 (1)
Sars-cov-2 test positive (Investigations) | 1 (1) | 0 (0)
Systemic lupus erythematosus disease activity index abnormal (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Calciphylaxis (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 6 (6) | 8 (8)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 14 (17) | 18 (18)
Coagulopathy (Blood and lymphatic system disorders) | 2 (2) | 4 (5)
Cardiac ventricular thrombosis (Cardiac disorders) | 1 (1) | 2 (2)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 3 (4) | 3 (3)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Gout (Metabolism and nutrition disorders) | 4 (4) | 4 (4)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 6 (6) | 7 (8)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 (2) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 11 (12) | 4 (4)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 3 (3) | 5 (5)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 9 (9) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 10 (10) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 7 (7) | 8 (12)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Ketosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Latent autoimmune diabetes in adults (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 9 (9) | 12 (12)
Marasmus (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 5 (5)
Metabolic syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 10 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4)
Axial spondyloarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cardiomegaly (Cardiac disorders) | 1 (1) | 1 (1)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Hypertrophic osteoarthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Immobilisation syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 7 (8) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Oligoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 9 (9) | 8 (9)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Cardiomyopathy alcoholic (Cardiac disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Spinal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Spinal synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 3 (3) | 3 (3)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 4 (4)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Adrenal gland cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cardiorenal syndrome (Cardiac disorders) | 1 (1) | 1 (1)
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adult t-cell lymphoma/leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Cardiovascular insufficiency (Cardiac disorders) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (5)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (3)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Chronic coronary syndrome (Cardiac disorders) | 3 (3) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 9 (9)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Diffuse large b-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Ductal adenocarcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Chronic left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Essential thrombocythaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Fallopian tube cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Follicular lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 1 (1) | 1 (1)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (2)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Intracranial meningioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Joint neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3)
Lung adenocarcinoma stage i (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 9 (9) | 14 (16)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 7 (7)
Lung squamous cell carcinoma stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lymphoplasmacytoid lymphoma/immunocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0)
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Mediastinum neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Myeloproliferative neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Non-small cell lung cancer stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 3 (3) | 2 (2)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Oesophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Oropharyngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 4 (4)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Frederick's syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Pleural mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 7 (7)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Refractory cytopenia with unilineage dysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Heart valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small cell lung cancer extensive stage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Soft tissue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Hypertensive cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Squamous cell carcinoma of the vulva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Triple negative breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour embolism (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour perforation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Uterine neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Waldenstrom's macroglobulinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 3 (4)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Bell's palsy (Nervous system disorders) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 1 (1) | 2 (2)
Brain stem infarction (Nervous system disorders) | 5 (5) | 1 (1)
Carotid artery occlusion (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 3 (3) | 1 (1)
Carotid artery thrombosis (Nervous system disorders) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (2)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 2 (2)
Left ventricular failure (Cardiac disorders) | 5 (5) | 8 (8)
Cerebral arteriosclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haematoma (Nervous system disorders) | 0 (0) | 2 (2)
Cerebral haemorrhage (Nervous system disorders) | 2 (2) | 4 (4)
Cerebral infarction (Nervous system disorders) | 11 (11) | 11 (11)
Cerebrovascular accident (Nervous system disorders) | 5 (5) | 3 (3)
Cerebrovascular disorder (Nervous system disorders) | 2 (2) | 0 (0)
Cervical cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 2 (2) | 1 (1)
Cubital tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Dementia alzheimer's type (Nervous system disorders) | 1 (1) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Microvascular coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 5 (5) | 3 (3)
Drop attacks (Nervous system disorders) | 1 (1) | 0 (0)
Embolic cerebral infarction (Nervous system disorders) | 1 (2) | 0 (0)
Embolic stroke (Nervous system disorders) | 7 (7) | 5 (5)
Encephalopathy (Nervous system disorders) | 0 (0) | 2 (2)
Epilepsy (Nervous system disorders) | 2 (2) | 3 (3)
Focal dyscognitive seizures (Nervous system disorders) | 1 (1) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 10 (10) | 9 (10)
Mitral valve calcification (Cardiac disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 3 (3) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial haematoma (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 70 (76) | 65 (70)
Lacunar infarction (Nervous system disorders) | 1 (1) | 3 (3)
Lacunar stroke (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 2 (2)
Mitral valve disease (Cardiac disorders) | 2 (2) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Myelopathy (Nervous system disorders) | 0 (0) | 1 (1)
Myoclonic epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Myoclonus (Nervous system disorders) | 1 (1) | 1 (1)
Myxoedema coma (Nervous system disorders) | 1 (1) | 0 (0)
Parkinson's disease (Nervous system disorders) | 0 (0) | 4 (4)
Parkinsonism (Nervous system disorders) | 1 (1) | 0 (0)
Partial seizures (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Polyneuropathy alcoholic (Nervous system disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 8 (9) | 6 (7)
Post stroke epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 4 (4) | 1 (1)
Quadriparesis (Nervous system disorders) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 5 (5) | 2 (2)
Spinal stroke (Nervous system disorders) | 1 (1) | 0 (0)
Spondylitic myelopathy (Nervous system disorders) | 0 (0) | 2 (2)
Status epilepticus (Nervous system disorders) | 2 (2) | 2 (2)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Mitral valve stenosis (Cardiac disorders) | 0 (0) | 3 (3)
Syncope (Nervous system disorders) | 18 (18) | 21 (21)
Thalamic infarction (Nervous system disorders) | 0 (0) | 1 (1)
Thrombotic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Thrombotic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 6 (7) | 5 (5)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Uraemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Vascular encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Myocardial fibrosis (Cardiac disorders) | 1 (1) | 0 (0)
Vertebrobasilar stroke (Nervous system disorders) | 0 (0) | 1 (1)
Device dislocation (Product Issues) | 0 (0) | 1 (1)
Device failure (Product Issues) | 2 (2) | 0 (0)
Device fastener issue (Product Issues) | 0 (0) | 1 (1)
Device malfunction (Product Issues) | 1 (1) | 1 (1)
Device occlusion (Product Issues) | 1 (1) | 0 (0)
Device power source issue (Product Issues) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 2 (2)
Completed suicide (Psychiatric disorders) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 15 (16) | 18 (19)
Confusional state (Psychiatric disorders) | 2 (4) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 2 (2)
Delirium tremens (Psychiatric disorders) | 1 (1) | 0 (0)
Delusion (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 1 (2) | 0 (0)
Mental status changes (Psychiatric disorders) | 2 (2) | 7 (9)
Organic brain syndrome (Psychiatric disorders) | 2 (2) | 1 (1)
Psychogenic respiratory distress (Psychiatric disorders) | 0 (0) | 1 (1)
Psychomotor retardation (Psychiatric disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 2 (2) | 4 (4)
Substance abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 54 (64) | 63 (78)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 12 (12) | 10 (12)
Cystitis glandularis (Renal and urinary disorders) | 1 (1) | 0 (0)
Cystitis haemorrhagic (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 4 (5) | 4 (7)
Myxomatous mitral valve degeneration (Cardiac disorders) | 0 (0) | 1 (1)
Glomerulonephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 5 (6) | 7 (7)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 3 (3)
Nephropathy toxic (Renal and urinary disorders) | 2 (2) | 2 (2)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 1 (1)
Obstructive nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Prerenal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal amyloidosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nodal rhythm (Cardiac disorders) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal cyst ruptured (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 9 (9) | 11 (11)
Renal haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 7 (7) | 7 (7)
Renal injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary fistula (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 2 (2) | 0 (0)
Evans syndrome (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Urinary tract inflammation (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 2 (2)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acquired phimosis (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 4 (4) | 3 (3)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Endometrial atrophy (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatomegaly (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 2 (2)
Scrotal ulcer (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vulvovaginal inflammation (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 6 (7)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 16 (19) | 17 (20)
Allergic respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 9 (11)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 21 (30) | 18 (26)
Chronic respiratory disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Right ventricular failure (Cardiac disorders) | 0 (0) | 2 (4)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (5)
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nocturnal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Platypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 7 (8)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sinoatrial block (Cardiac disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 9 (9)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary hilum mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 5 (5)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 17 (19)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 3 (5) | 6 (8)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 9 (9) | 11 (11)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (5)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cardiac assistance device user (Social circumstances) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 3 (3) | 1 (1)
Aortic aneurysm rupture (Vascular disorders) | 0 (0) | 1 (1)
Aortic dissection (Vascular disorders) | 1 (1) | 1 (1)
Aortic stenosis (Vascular disorders) | 4 (4) | 5 (5)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Bleeding varicose vein (Vascular disorders) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 1 (1)
Extremity necrosis (Vascular disorders) | 0 (0) | 2 (2)
Femoral artery aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Femoral artery embolism (Vascular disorders) | 0 (0) | 1 (1)
Haematocoele (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 2 (2) | 3 (3)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 14 (16) | 9 (10)
Supraventricular tachycardia (Cardiac disorders) | 2 (2) | 2 (3)
Hypertensive crisis (Vascular disorders) | 3 (3) | 1 (1)
Hypertensive emergency (Vascular disorders) | 1 (1) | 1 (1)
Hypertensive urgency (Vascular disorders) | 4 (4) | 3 (3)
Hypotension (Vascular disorders) | 10 (10) | 6 (6)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1)
Iliac artery stenosis (Vascular disorders) | 0 (0) | 1 (1)
Lymphoedema (Vascular disorders) | 2 (2) | 0 (0)
Malignant hypertension (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 3 (3) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 24 (24) | 18 (21)
Tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Peripheral artery aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 4 (4) | 3 (3)
Peripheral artery stenosis (Vascular disorders) | 2 (2) | 2 (2)
Peripheral artery thrombosis (Vascular disorders) | 2 (2) | 1 (1)
Peripheral embolism (Vascular disorders) | 2 (2) | 2 (2)
Peripheral ischaemia (Vascular disorders) | 5 (7) | 9 (12)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 2 (2) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 2 (2)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Varicose ulceration (Vascular disorders) | 1 (1) | 0 (0)
Varicose vein (Vascular disorders) | 1 (1) | 0 (0)
Vascular insufficiency (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1)
Vessel perforation (Vascular disorders) | 1 (1) | 0 (0)
Tachycardia induced cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Torsade de pointes (Cardiac disorders) | 2 (2) | 0 (0)
Trifascicular block (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 6 (6) | 6 (6)
Ventricular tachycardia (Cardiac disorders) | 13 (15) | 13 (16)
Congenital hypercoagulation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Retinal arteriovenous malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapa 10 mg (N=3126) | Placebo (N=3127)
Atrial fibrillation (Cardiac disorders) | 86 (103) | 61 (70)
Urinary tract infection (Infections and infestations) | 113 (142) | 112 (128)
Cardiac failure (Cardiac disorders) | 179 (240) | 214 (255)
Hypertension (Vascular disorders) | 84 (104) | 102 (136)
Hypotension (Vascular disorders) | 69 (80) | 61 (68)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-11-12): https://cdn.clinicaltrials.gov/large-docs/13/NCT03619213/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-08): https://cdn.clinicaltrials.gov/large-docs/13/NCT03619213/SAP_001.pdf